CLINICAL TRIAL: NCT05489315
Title: Quantifying the Impact of the Peanut Ball on the Duration of the Active Stage of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Rachel Nelson, Co-Principal Investigator, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-08072-FB
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Labor Onset and Length Abnormalities; Prolonged Labor; Labor Long; Labor; Poor
Keywords: peanut ball; labor; cesarean section
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Positioning (Other): Participants who are randomly assigned to NOT receive a peanut ball will undergo placement on a wedge pillow and/or traditional positioning during their labor progression at 6cm cervical dilation.
  Interventions: Other: Traditional positioning
- Peanut Ball Positioning (Experimental): Participants who are randomly assigned to receive a peanut ball will be positioned with a peanut ball at 6cm cervical dilation.
  Interventions: Device: Positioning with peanut ball

INTERVENTIONS:
Device: Positioning with peanut ball — If participants are randomly selected to receive a peanut ball, the intent is for the patient to remain on the peanut ball during their labor progression.
  Arms: Peanut Ball Positioning
Other: Traditional positioning — If participants are randomly selected to NOT receive a peanut ball, the intent is for the patient to undergo traditional positioning/use wedge pillows during their labor progression.
  Arms: Traditional Positioning

SUMMARY:
Prolonged labor is associated with adverse maternal and fetal outcomes including infection, postpartum hemorrhage and increased NICU admission. One of the most common indications for cesarean section in the US is prolonged labor. Maternal positioning through labor facilitated by birthing balls is believed to help facilitate labor. Current data is inconclusive on whether or not the use of birthing balls is advantageous in a statistically significant manner.

In this prospective randomized controlled trial, participants will be randomly selected to receive either the experimental intervention (repositioning peanut ball during labor) or the control intervention (the standard therapy of traditional repositioning during labor).

Primary outcome: Time of active labor to delivery with and without use of the peanut ball.

Secondary outcome: Cesarean section frequency.

ELIGIBILITY:
Inclusion Criteria:

* Fetus must be vertex in position at the time of admission to L&D
* Pregnant patients age 16 years old and above
* Singleton pregnancy (ie. one fetus)
* Patients who receive induction and augmentation of labor may be included
* Include both nulliparous and multiparous women
* Patients with HTN, diabetes, and obesity at any point in their pregnancy may be included
* Patients may be included in the study regardless of whether or not they received an epidural
* Patients who have been randomly assigned to receive a peanut ball must be placed on the peanut ball at 6cm dilation, not earlier.
* Patients who present to L&D dilated to 4cm may be included

Exclusion Criteria:

* TOLACs and VBACs will be excluded
* Multiple gestation will be excluded
* Category 3 fetal tracing will be excluded
* Chorioamnionitis will be excluded
* Patients who present to L&D at 6cm cervical dilation will be excluded
* Patients placed on the peanut ball before 6cm cervical dilation will be excluded
* Patients with fetal malpresentation will be excluded

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-05-19 (Estimated); Study Completion 2023-05-19 (Estimated)

PRIMARY OUTCOMES:
Rate of active stage of labor | Expected <6 hours
  Length of time from progression of 6cm cervical dilation to 10cm

SECONDARY OUTCOMES:
Cesarean section rate | < 48 hours
  Proportion of patients who undergo delivery by cesarean section

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Regional One Health Outpatient Center, Memphis, Tennessee
  - Regional One Health, Memphis, Tennessee
  - Regional One Health - Hollywood Clinic, Memphis, Tennessee
  - Regional One Health - Kirby Primary Care Clinic, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tussey CM, Botsios E, Gerkin RD, Kelly LA, Gamez J, Mensik J. Reducing Length of Labor and Cesarean Surgery Rate Using a Peanut Ball for Women Laboring With an Epidural. J Perinat Educ. 2015;24(1):16-24. doi: 10.1891/1058-1243.24.1.16. PMID 26937158
- [Background] Roth C, Dent SA, Parfitt SE, Hering SL, Bay RC. Randomized Controlled Trial of Use of the Peanut Ball During Labor. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):140-6. doi: 10.1097/NMC.0000000000000232. PMID 26859467
- [Background] Mercier RJ, Kwan M. Impact of Peanut Ball Device on the Duration of Active Labor: A Randomized Control Trial. Am J Perinatol. 2018 Aug;35(10):1006-1011. doi: 10.1055/s-0038-1636531. Epub 2018 Mar 6. PMID 29510425
- [Background] Grenvik JM, Rosenthal E, Saccone G, Della Corte L, Quist-Nelson J, Gerkin RD, Gimovsky AC, Kwan M, Mercier R, Berghella V. Peanut ball for decreasing length of labor: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2019 Nov;242:159-165. doi: 10.1016/j.ejogrb.2019.09.018. Epub 2019 Sep 20. PMID 31600716

DOCUMENTS (1):
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT05489315/ICF_000.pdf